CLINICAL TRIAL: NCT01913613
Title: REDUCE LAP-HF TRIAL: A Study to Evaluate the DC Devices, Inc. IASD™ System II to REDUCE Elevated Left Atrial Pressure in Patients With Heart Failure
Brief Title: REDUCE LAP-HF TRIAL
Acronym: REDUCE LAP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-01
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the IASD device
  Interventions: Device: IASD

INTERVENTIONS:
Device: IASD — IASD device implantation

SUMMARY:
The objective of this clinical study is to evaluate the safety and performance of the IASD System II in the treatment of heart failure patients with elevated left atrial pressure, who remain symptomatic despite appropriate medical management.

ELIGIBILITY:
Key Inclusion Criteria:

1. Chronic symptomatic Heart Failure (HF) documented by one or more of the following:

   1. New York Heart Association (NYHA) Class II/III/ambulatory class IV symptoms (Paroxysmal nocturnal dyspnea, Orthopnea, Dyspnea on mild or moderate exertion) at screening visit; or signs (Any rales post cough, Chest x-ray demonstrating pulmonary congestion,) within past 12 months;
   2. One hospital admission for which HF was a major component of the hospitalization within the 12 months prior to study entry (transient heart failure in the context of myocardial infarction does not qualify);
   3. On-going management with recommended heart failure medications and comorbidities for several months according to the guidelines (2012 ESC Guidelines for diagnosis and Treatment of Acute and Chronic Heart Failure).
2. Age ≥ 40 years old
3. Left ventricular ejection fraction (obtained by echocardiography) ≥ 40%
4. Elevated left ventricular filling pressures with a gradient compared to CVP documented by :

   1. PCWP or LVEDP at rest ≥ 15 mmHg, and greater than CVP, OR
   2. PCWP during supine bike exercise ≥ 25mm Hg, and CVP < 20 mm Hg

Key Exclusion Criteria:

3. Severe heart failure defined as:

1. ACC/AHA/ESC Stage D heart failure, Non-ambulatory NYHA Class IV HF;
2. Fick Cardiac Index < 2.0 L/min/m2
3. Requiring inotropic infusion (continuous or intermittent) within the past 6 months
4. Patient is on the cardiac transplant waiting list 4. Inability to perform 6 Minute Walk Test 5. Known significant coronary artery disease (stenosis >70%) 6. History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months 7. Known severe carotid artery stenosis (> 70%) 8. Presence of significant valve disease defined by echocardiography as: a) Mitral valve regurgitation defined as grade >2+ MR b) Tricuspid valve regurgitation defined as grade ≥ 2+ TR; c) Aortic valve disease defined as ≥ 2+ AR or moderate AS

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
MACCE | 6 months
  subjects who experience major adverse cardiac and cerebrovascular events (MACCE) defined as death, stroke, MI; or subjects who experience a systemic embolic event (excluding pulmonary thromboembolism)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Komtebedde, DVM, Study Chair — Corvia Medical
Locations (26):
- Australia (3):
  - The Prince Charles Hospital, Brisbane
  - David Kaye, Melbourne
  - St. Vincent Hospital, Sydney
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Allgemeines Krankenhaus Univesitäts Kliniken, Vienna
- OLVZ Aalst, Aalst, Belgium
- Homolka Hospital, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - CHRU de Lille, Lille
  - CHU de Nantes, Nantes
  - Hôpital Bichat, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Rangueil, Toulouse
- Germany (7):
  - Universitatklinikum Duseldorf, Düsseldorf
  - Georg-August-Universitat, Göttingen
  - Asklepios Klinik St George, Hamburg
  - Cardiologicum CRC, Hamburg
  - University of Heidelberg, Heidelberg
  - Universtitaät Kliniku Schlewig Holstein, Kiel
  - Klinikum der Universität Munchen, Munich
- St Antonius Ziekenhuis, Nieuwegein, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Fourth Military Hospital, Wroclaw, Poland
- United Kingdom (3):
  - Golden Jubilee Hospital, Glasgow
  - Royal Brompton/Harefield Trust, Harefield
  - King's College, London

REFERENCES:
- [Background] Hasenfuss G, Gustafsson F, Kaye D, Shah SJ, Burkhoff D, Reymond MC, Komtebedde J, Hunlich M; Reduce LAP-HF Trial Investigators. Rationale and Design of the Reduce Elevated Left Atrial Pressure in Patients With Heart Failure (Reduce LAP-HF) Trial. J Card Fail. 2015 Jul;21(7):594-600. doi: 10.1016/j.cardfail.2015.05.008. Epub 2015 Jun 6. PMID 26055211
- [Result] Hasenfuss G, Hayward C, Burkhoff D, Silvestry FE, McKenzie S, Gustafsson F, Malek F, Van der Heyden J, Lang I, Petrie MC, Cleland JG, Leon M, Kaye DM; REDUCE LAP-HF study investigators. A transcatheter intracardiac shunt device for heart failure with preserved ejection fraction (REDUCE LAP-HF): a multicentre, open-label, single-arm, phase 1 trial. Lancet. 2016 Mar 26;387(10025):1298-304. doi: 10.1016/S0140-6736(16)00704-2. PMID 27025436
- [Result] Kaye DM, Hasenfuss G, Neuzil P, Post MC, Doughty R, Trochu JN, Kolodziej A, Westenfeld R, Penicka M, Rosenberg M, Walton A, Muller D, Walters D, Hausleiter J, Raake P, Petrie MC, Bergmann M, Jondeau G, Feldman T, Veldhuisen DJ, Ponikowski P, Silvestry FE, Burkhoff D, Hayward C. One-Year Outcomes After Transcatheter Insertion of an Interatrial Shunt Device for the Management of Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2016 Dec;9(12):e003662. doi: 10.1161/CIRCHEARTFAILURE.116.003662. PMID 27852653
- [Result] Wolsk E, Kaye D, Borlaug BA, Burkhoff D, Kitzman DW, Komtebedde J, Lam CSP, Ponikowski P, Shah SJ, Gustafsson F. Resting and exercise haemodynamics in relation to six-minute walk test in patients with heart failure and preserved ejection fraction. Eur J Heart Fail. 2018 Apr;20(4):715-722. doi: 10.1002/ejhf.976. Epub 2017 Sep 26. PMID 28949052
- [Result] Kaye DM, Petrie MC, McKenzie S, Hasenfubeta G, Malek F, Post M, Doughty RN, Trochu JN, Gustafsson F, Lang I, Kolodziej A, Westenfeld R, Penicka M, Rosenberg M, Hausleiter J, Raake P, Jondeau G, Bergmann MW, Spelman T, Aytug H, Ponikowski P, Hayward C; REDUCE LAP-HF study investigators. Impact of an interatrial shunt device on survival and heart failure hospitalization in patients with preserved ejection fraction. ESC Heart Fail. 2019 Feb;6(1):62-69. doi: 10.1002/ehf2.12350. Epub 2018 Oct 11. PMID 30311437
- [Result] Wessler J, Kaye D, Gustafsson F, Petrie MC, Hasenfubeta G, Lam CSP, Borlaug BA, Komtebedde J, Feldman T, Shah SJ, Burkhoff D; REDUCE-LAP-HF Trial Investigators and Advisors. Impact of Baseline Hemodynamics on the Effects of a Transcatheter Interatrial Shunt Device in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2018 Aug;11(8):e004540. doi: 10.1161/CIRCHEARTFAILURE.117.004540. PMID 30354556
- [Result] Hanff TC, Kaye DM, Hayward CS, Post MC, Malek F, Hasenfubeta G, Gustafsson F, Burkhoff D, Shah SJ, Litwin SE, Kahwash R, Hummel SL, Borlaug BA, Solomon SD, Lam CSP, Komtebedde J, Silvestry FE; REDUCE LAP-HF study investigators, and research staff. Assessment of Predictors of Left Atrial Volume Response to a Transcatheter InterAtrial Shunt Device (from the REDUCE LAP-HF Trial). Am J Cardiol. 2019 Dec 15;124(12):1912-1917. doi: 10.1016/j.amjcard.2019.09.019. Epub 2019 Sep 26. PMID 31653352
- [Derived] Obokata M, Reddy YNV, Shah SJ, Kaye DM, Gustafsson F, Hasenfubeta G, Hoendermis E, Litwin SE, Komtebedde J, Lam C, Burkhoff D, Borlaug BA. Effects of Interatrial Shunt on Pulmonary Vascular Function in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2019 Nov 26;74(21):2539-2550. doi: 10.1016/j.jacc.2019.08.1062. PMID 31753198